CLINICAL TRIAL: NCT03619577
Title: The Effectiveness of Combining Physical Exercise and Cognitive Training for Individuals With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201711EM006
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; cognitive training; exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential training-high frequency (Experimental): The participants of HF will receive a total of 36 training sessions, and each session will contain 90-105 minutes of training. The participants in this group will first perform 45-55 minutes of physical exercise followed by 45-50 minutes of cognitive training. The participants in this group participate in multimodel exercise programs including aerobic exercise, balance, and strength training. The entire program will contain 5-10 minutes of warm-up, 35-40 minutes of physical exercise, and 5 minutes of cool-down. Then, the participants will practice tasks that involve the abilities of visuospatial processing, attention, memory, language, and/or executive functions for 45-50 minutes.
  Interventions: Behavioral: Sequential training
- Sequential training-low frequency (Experimental): The participants of LF will receive a total of 12 training sessions, and each session will contain 90-105 minutes of training. The participants in this group will first perform 45-55 minutes of physical exercise followed by 45-50 minutes of cognitive training. The participants in this group participate in multimodel exercise programs including aerobic exercise, balance, and strength training. The entire program will contain 5-10 minutes of warm-up, 35-40 minutes of physical exercise, and 5 minutes of cool-down. Then, the participants will practice tasks that involve the abilities of visuospatial processing, attention, memory, language, and/or executive functions for 45-50 minutes.
  Interventions: Behavioral: Sequential training

INTERVENTIONS:
Behavioral: Sequential training — For cognitive training, the BrainHQ program, self-made teaching aids and board games will be used to train different cognitive functions of the participants. For physical exercise, we design the programs that involve balance or strength training components in the aerobic exercises. All participants will first perform 60 minutes of physical exercise followed by 60 minutes of cognitive training.

SUMMARY:
Mild cognitive impairment (MCI) is a syndrome defined as an intermediate stage between cognitively intact and clinically diagnosed dementia. The progression rate from MCI to dementia ranges from 10 to 15% each year, resulting in increased family care and medical expenses. Therefore, providing effective interventions are necessary. Combining cognitive training and physical exercise training appears to have effects to prevent the progression of MCI to Alzheimer's disease or other severe cognitive impairment. It was proposed that cognitively challenging stimulations can increase the neural network and promote neural plasticity, which are essential for preventing cognitive decline in patients with MCI. The studies also showed that physical exercise induces positive effects on cerebral blood flow and induces brain activation changes of the frontal, parietal, and temporal areas; these cortical areas are especially important for memory and other cognitive functions. However, it is yet not clear the appropriate frequency of the effective intervention for patients with MCI. Thus, this study aims to compare the intervention effects of high frequency sequential and low frequency sequential training for patients with MCI.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is a syndrome defined as an intermediate stage between cognitively intact and clinically diagnosed dementia. The progression rate from MCI to dementia ranges from 10 to 15% each year, resulting in increased family care and medical expenses. Therefore, providing effective interventions are necessary. Combining cognitive training and physical exercise training appears to have effects to prevent the progression of MCI to Alzheimer's disease or other severe cognitive impairment. It was proposed that cognitively challenging stimulations can increase the neural network and promote neural plasticity, which are essential for preventing cognitive decline in patients with MCI. The studies also showed that physical exercise induces positive effects on cerebral blood flow and induces brain activation changes of the frontal, parietal, and temporal areas; these cortical areas are especially important for memory and other cognitive functions. However, it is yet not clear the appropriate frequency of the effective intervention for patients with MCI. Thus, this study aims to compare the intervention effects of high frequency sequential and low frequency sequential training for patients with MCI.

Investigators anticipate recruiting a total of 80 participants with MCI. The participants will be assigned into 2 groups: high frequency sequential training (HF) and low frequency sequential training (LF) groups. The participants of HF will receive a total of 36 training sessions, and each session will contain 90-105 minutes of training. The participants of LF will receive a total of 12 training sessions, and each session will contain 90-105 minutes of training. The BrainHQ program, self-made teaching aids and board games will be used to train different cognitive functions of the participants. For physical exercise, Investigators design the programs that involve balance or strength training components in the aerobic exercises. All participants will first perform 45-55 minutes of physical exercise followed by 45-50 minutes of cognitive training. Investigators plan to assess the participants before and after the intervention programs. The primary outcome measures are cognitive functions, including visuospatial processing, attention, memory, and/or executive functions. The secondary outcome measures include physical functions and activities of daily living (ADLs). Investigators expect to use the paired-t test and analysis of covariance (ANCOVA) to analyze differences in baseline characteristics and baseline outcome measures between the groups and determine the intervention effect for the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* able to follow instruction (MMSE>= 17)
* self- or informant-reported memory or cognitive complaint.

Exclusion Criteria:

* recent myocardial infarction,heart failure,recent heart surgery,
* severe asthma, concomitant with other neurological disorders, or joint deformity that might prevents them performing exercise or cognitive training.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA) | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Change scores of the Stroop test | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The Stroop test will be used to assess the processing speed, inhibition, set-shifting, and selective attention abilities. The participants will be tested under 2 conditions: congruent and incongruent conditions. In the congruent condition, the color ink of a word is consistent with the written color name; while the color ink differs from the written color name under the incongruent condition.
Change scores of the Dual-task test | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically
Change scores of the Timed up and go (TUG) test | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The TUG test will be used to assess the mobility and dynamic balance ability. The participants will be required to stand up from a chair, walk 3 meters, turn around, then walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers and frail elderly (Podsiadlo & Richardson, 1991). The test-retest reliability of TUG on individuals with cognitive impairment was excellent.
Change scores of the Wechsler Memory Scale (WMS) | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  Tests of the Wechsler Memory Scale (WMS) will be used to measure the memory functions of an individual. The WMS have high reliability and validity, and is often used to differentiate individuals with memory deficits and those with intact cognitive functions. In addition, WMS could be used to assess cognitive improvements after an intervention or treatment. There are eight Primary Indexes (Auditory Immediate (was Verbal), Visual Immediate (was Visual), Immediate Memory (new), Auditory Delayed (new), Visual Delayed (new), Auditory Reception Delayed (new), General Memory (only delayed subtest scores), and Working Memory), which constitute Immediate Memory, General (Delayed) Memory, and Working Memory (was Attention/Concentration). Approximately 60 to 90 minutes is required for completion.
Change scores of the Lawton Instrumental Activities of Daily Living Scale (IADL) | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  Assess activities of daily living. There are 8 domains of function measured with the Lawton IADL scale, including ability to use phone,shopping, food preparation, housekeeping, laundering, mode of transportation, responsibility for own medications,and ability to handle finances. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent). For each category, circle the item description that most closely resembles the client's highest functional level (either 0 or 1).
Change scores of the Wechsler Adult Intelligence Scale (WAIS) | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  Subtests of the Wechsler Adult Intelligence Scale (WAIS) will be used to measure the cognitive functions of an individual. The WAIS have high reliability and validity, and is often used to differentiate individuals with cognitive deficits and those with intact cognitive functions. In addition, WAIS could be used to assess cognitive improvements after an intervention or treatment.
Change scores of Memory complaint questionnaire | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The MAC-Q consists of six items. The first five items relate to specific situations that are frequently reported as troublesome for those with declining memory, and the last item broadly measures overall self-perceived memory decline. Respondents must choose one of the 5 options ranging from much better now to much worse now. The total possible score is 30 points.
Change scores of Spatial Span Test | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The Spatial Span Task is a behavioral measure of working memory capacity, the cognitive ability to store and manage information on a transient basis.
  On each trial the squares change from white to a different color in a sequence with variable orders and colors. The task exists with two variants: forward-span and backward-span. In the forward-span variant, at the end of each list participants attempt to recall the squares in the order they changed color by typing keys corresponding to each square via keypress. In the backward-span variant, at the end of each list participants attempt to recall the squares in the reverse order that they changed color. The difficulty level is systematically increased by varying the number of boxes on each trial from two boxes (easiest) to nine boxes (most difficult).

SECONDARY OUTCOMES:
Change scores of the short form of the Geriatric Depression Scale (GDS-SF) | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The Chinese version of short form GDS will be used. The short-form version comprising 15 items. Answers indicating depression are in bold and italicized; score one point for each one selected. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
Change scores of the Community Integration Questionnaire (CIQ) | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  The CIQ measures items relevant to home integration, social integration, and productive activities.
Change scores of the Everyday Cognition scales (ECog)-12 items | baseline, posttest (around 12 weeks after baseline), follow-up (6 months after completing intervention sessions)
  To detect cognitive and functional decline. The ECog shows promise as a useful tool for the measurement of general and domain-specific everyday functions in the elderly. There are six domains (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided Attention) in ECog. Lower scores represent a higher level of function in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chuang IC, Chen IC, Wu YR, Li KY. Prediction and mediation analysis for treatment responses to combined cognitive and physical training for older adults. Sci Rep. 2024 May 8;14(1):10571. doi: 10.1038/s41598-024-61407-6. PMID 38720025
- [Derived] Chuang IC, Chen IC, Su KH, Wu YR, Wu CY. The effects of high versus low frequency of combined physical and cognitive training on cognitive function in older adults with cognitive decline: a quasi-experimental study. BMC Geriatr. 2023 Feb 14;23(1):94. doi: 10.1186/s12877-023-03802-8. PMID 36788482